CLINICAL TRIAL: NCT01712789
Title: A Multicenter, Single-arm, Open-label Study With Pomalidomide in Combination With Low Dose Dexamethasone in Subjects With Refractory or Relapsed and Refractory Multiple Myeloma
Brief Title: Evaluation of Safety of Pomalidomide in Combination With Dexamethasone (Low Dose) in Patients With Refractory or Relapsed and Refractory Multiple Myeloma
Acronym: STRATUS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-4047-MM-010; 2012-001888-78 (EudraCT Number)
Record Dates: First submitted 2012-10-22; First posted 2012-10-24 (Estimated); Results first posted 2022-01-10 (Actual); Last update posted 2022-01-10 (Actual); Status verified 2021-12

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Relapsed Multiple Myeloma; Relapsed and refractory Multiple Myeloma; Pomalidomide; Dexamethasone
MeSH Terms: conditions — Multiple Myeloma; Recurrence | interventions — pomalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pomalidomide plus Dexamethasone (Experimental): Pomalidomide 4mg by mouth (PO) daily days 1 through 21 of a 28 day cycle and dexamethasone 40mg/day PO for those ≤75 years of age or 20mg/day for those greater than 75 years of age on Days 1, 8, 15 and 22 of a 28 day cycle.
  Interventions: Drug: Pomalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Pomalidomide — Oral Pomalidomide at the starting dose of 4 mg on Days 1-21 of a 28-day cycle
Drug: Dexamethasone — Oral Low dose Dexamethasone at the starting dose of 40mg/day (≤ 75 years old) or 20 mg/day (> 75 years old) on Days 1, 8, 15 and 22 of a 28-day cycle.

SUMMARY:
The primary purpose of the study is to evaluate the safety and efficacy and to generate PK and biomarker data for the combination of pomalidomide and low-dose dexamethasone in patients with refractory or relapsed and refractory multiple myeloma.

The study consists of a Screening phase within 28 days prior to cycle 1 day 1, a Treatment phase and a Follow-up phase which starts within 28 days of discontinuation from study treatment, every 3 months for up to 5 years.

In addition, the collection of steady-state PK data from a large population will enable robust population PK and assess Pomalidomide exposure response analyses.

The exploratory objectives of the study are to investigate potential markers predictive of POM response or resistance and pharmacodynamic markers.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years old, who must understand and voluntarily sign an Informed Consent.
* Patients must have documented diagnosis of Multiple Myeloma and have measurable disease.
* Patients must have undergone prior treatment with ≥ 2 treatments lines, of anti-myeloma therapy.
* Patients must have either refractory or relapsed and refractory disease.
* Patients must have received at least 2 consecutive cycles of prior treatment that include lenalidomide and bortezomib, either alone or in combination regimens.
* Patients must have received adequate alkylator therapy

Exclusion Criteria:

* Prior history of malignancies, other than Multiple Myeloma.
* Previous therapy with Pomalidomide, hypersensitivity to thalidomide and lenalidomide or dexamethasone.
* Patients who received an allogeneic bone marrow or allogeneic peripheral blood stem cell transplant.
* Patients who are planning for or who are eligible for stem cell transplant.
* Patients who received major surgery and any anti-myeloma drug therapy within the last 14 days of starting study treatment.
* Patients with a current disease that can interfere with protocol procedures or study treatment.
* Patients unable or unwilling to undergo antithrombotic prophylactic treatment.
* Pregnant or breastfeeding females.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 682 (Actual)
Dates: Start 2012-11-06 (Actual); Primary Completion 2019-12-11 (Actual); Study Completion 2019-12-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Peluso, MBBS, DCPSA, Study Director — Bristol-Myers Squibb
Locations (112):
- Austria (4):
  - Medical University of Graz, Graz
  - Medizinische Universitat Innsbruck, Innsbruck
  - Wilhelminenspital Vienna, Vienna
  - Medical University of Vienna, Vienna
- Belgium (7):
  - AZ St-Jan Brugge Oostende AV, Bruges
  - Institut Jules Bordet, Brussels
  - VUB Vrije Universiteit Brussel, Brussels
  - UZ Gent, Ghent
  - UZ Leuven, Leuven
  - Centre Hospitalier Universitaire de Liege, Liège
  - CHU Mont -Godinne, Yvoir
- Denmark (3):
  - Aarhus University Hospital, Aarhus
  - Odense University Hospital, Odense
  - Vejle Hospital, Vejle
- Tartu University Hospital Clinic, Tartu, Estonia
- Finland (2):
  - Helsingin yliopistollinen keskussairaala, Helsinki
  - Turku University Hospital, Turku
- France (13):
  - Centre Hospitalier de la cote basque, Bayonne
  - Hopital Henri Mondor, Créteil
  - Hopital A. Michallon, La Tronche
  - CHRU Claude Huriez, Lille
  - Institut Paoli Calmette Hematologie, Marseille
  - CHU Hotel Dieu, Nantes
  - Hopital Saint Antoine, Paris
  - Service Hemato-Immunologie Hopital St Louis, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - CHU de Reims, Reims
  - Hematologie - CHU Purpan, Toulouse
  - CHRU Hopital Bretonneau, Tours
  - CHU Nancy Hematology, Vandœuvre-lès-Nancy
- Germany (17):
  - Charite, Campus Benjamin Franklin Universitatsmedizin Berlin, Berlin
  - Klinikum Chemnitz, Chemnitz
  - Klinikum der Universitat zu Koln, Cologne
  - Universitatsklinikum Carl Gustav Carus, Dresden
  - Universitatsklinkikum DusseldorfKlinik fur Hamatologie, Onkologie und klin. Immunoligie, Düsseldorf
  - Universitatsklinikum Essen-, Essen
  - Universitatsklinikum Freiburg Medizinische Klinik und Poliklinik, Freiburg im Breisgau
  - Abt Haematologie - Onkologie / Allg. Krankenhaus Altona, Hamburg
  - Universitatsklinikum Heidelberg, Heidelberg
  - Universitatsklinikum Jena, Jena
  - University of Schleswig Holstein, Kiel
  - Universitatsklinikum Leipzig, Leipzig
  - TU München - Klinikum rechts der Isar, München
  - Universitatsklinik MuensterMedizinische Klinik A, Münster
  - UKT Universitaetsklinikum Tuebingen, Tübingen
  - University Hospital of Ulm, Ulm
  - Universitatsklinikum Wurzburg, Würzburg
- University of Athens, Athens, Greece
- Ireland (3):
  - Cork University HospitalHaematology Consultant, Wilton, Cork
  - Mater Misericordiae University Hospital, Dublin
  - University Hospital Galway, Galway
- Italy (15):
  - Ospedali Riuniti di Ancona, Ancona
  - A.O. Policlinico - Università di Bari, Bari
  - University of Bologna, Bologna
  - Ospedale Ferrarotto, Catania
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - ASST Grande Ospedale Metropolitano Niguarda, Milano, Milan
  - Universita degli Studi di Padova, Padua
  - Casa di Cura La Maddalena, Palermo
  - Ospedale Civile di Piacenza, Piacenza
  - Azienda Ospedaliero-Universitaria Pisana, Pisa
  - Universita degli Studi di Roma La Sapienza - Azienda Policlinico Umberto I, Roma
  - Ospedale Sant'Eugenio, Rome
  - Azienda Ospedaliera San Giovanni Battista - Ospedale Molinette, Torino
  - Azienda Ospedaliero-Universitaria Santa Maria della Misericordia die Udine, Udine
  - Ospedale San Bortolo, Vicenza
- Netherlands (5):
  - VU University Medical Center VU Medisch Centrum, Amsterdam
  - Universitair Medisch Centrum Groningen, Groningen
  - Erasmus Medical Center, Rotterdam
  - Haga Hospital, The Hague
  - University Medical Center Utrecht, Utrecht
- Norway (2):
  - Oslo University Hospital, Rikshospitalet HF, Oslo
  - St. Olavs Hospital Trondheim, Trondheim
- Poland (3):
  - Akademia Medyczna w Gdansku Katedra i Klinika Hematologii i Transplantologii, Gdansk
  - Szpitala Uniwersyteckiego w. Krakowie, Krakow
  - Instytut Hematologii i Transfuzjologii w Warszawie, Warsaw
- Portugal (4):
  - Hospital Universitario de Coimbra- Hospitais de Universidade de Coimbra, Coimbra
  - Instituto Portugues de Oncologia de Lisboa, Lisbon
  - Hospital de Santa Maria, Lisbon
  - Hospital Geral de Santo António - Serviço de Hematologia Clínica, Porto
- University Hospital Bratislava - Hospital Ss Cyril and Methodius, Bratislava, Slovakia
- Spain (15):
  - Hospital Universitari Germans Trias i Pujol, Badalona (Barcelona)
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario de Canarias, La Laguna (Tenerife)
  - Hospital de La Princesa, Madrid
  - Hospital Ramon y Cajal, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital 12 de Octubre, Madrid
  - Hospital Universitario Virgen De La Victoria, Málaga
  - Hospital Morales Meseguer, Murcia
  - Clinica Universidad de Navarra, Pamplona
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital de Donosti, San Sebastián (Guipuzcoa)
  - Hospital Clinico Universitario De Santiago De Compostela, Santiago de Compostela
  - Hospital Virgen de la Salud, Toledo
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia
- Sweden (2):
  - Universitetssjukhuset i Lund, Lund
  - Karolinska University HospitalSolna, Stockholm
- Switzerland (3):
  - Universitatsspital Bern, Bern
  - Hopitaux Universitaires de Geneve-HUG, Genèva
  - University Hospital Zurich, Zurich
- Turkey (Türkiye) (2):
  - Ankara University Medical Faculty Cebeci Hospital, Ankara
  - Ege University Medical School, Izmir
- United Kingdom (9):
  - Belfast City Hospital Haematology Department, Belfast Northern Ireland
  - Kent and Canterbury Hospital, Canterbury/Kent
  - Leeds Teaching Hospitals Trust, Leeds
  - Royal Liverpool University Hospital, Liverpool
  - Christie Hospital NHS Foundation Trust, Manchester
  - Newcastle Hospital Foundation Trust, Newcastle upon Tyne
  - Royal Marsden Hospital, Sutton (Surrey)
  - Southmead Hospital, Westbury-on-Trym/ Bristol
  - New Cross Hospital, Wolverhampton

REFERENCES:
- [Background] Dimopoulos MA, Palumbo A, Corradini P, Cavo M, Delforge M, Di Raimondo F, Weisel KC, Oriol A, Hansson M, Vacca A, Blanchard MJ, Goldschmidt H, Doyen C, Kaiser M, Petrini M, Anttila P, Cafro AM, Raymakers R, San-Miguel J, de Arriba F, Knop S, Rollig C, Ocio EM, Morgan G, Miller N, Simcock M, Peluso T, Herring J, Sternas L, Zaki MH, Moreau P. Safety and efficacy of pomalidomide plus low-dose dexamethasone in STRATUS (MM-010): a phase 3b study in refractory multiple myeloma. Blood. 2016 Jul 28;128(4):497-503. doi: 10.1182/blood-2016-02-700872. Epub 2016 May 25. PMID 27226434
- [Background] Moreau P, Dimopoulos MA, Richardson PG, Siegel DS, Cavo M, Corradini P, Weisel K, Delforge M, O'Gorman P, Song K, Chen C, Bahlis N, Oriol A, Hansson M, Kaiser M, Anttila P, Raymakers R, Joao C, Cook G, Sternas L, Biyukov T, Slaughter A, Hong K, Herring J, Yu X, Zaki M, San-Miguel J. Adverse event management in patients with relapsed and refractory multiple myeloma taking pomalidomide plus low-dose dexamethasone: A pooled analysis. Eur J Haematol. 2017 Sep;99(3):199-206. doi: 10.1111/ejh.12903. Epub 2017 Jun 14. PMID 28504846
- [Background] Qian X, Dimopoulos MA, Amatangelo M, Bjorklund C, Towfic F, Flynt E, Weisel KC, Ocio EM, Yu X, Peluso T, Sternas L, Zaki M, Moreau P, Thakurta A. Cereblon gene expression and correlation with clinical outcomes in patients with relapsed/refractory multiple myeloma treated with pomalidomide: an analysis of STRATUS. Leuk Lymphoma. 2019 Feb;60(2):462-470. doi: 10.1080/10428194.2018.1485915. Epub 2018 Aug 2. PMID 30068263
- [Background] Siegel DS, Weisel KC, Dimopoulos MA, Baz R, Richardson P, Delforge M, Song KW, San Miguel JF, Moreau P, Goldschmidt H, Cavo M, Jagannath S, Yu X, Hong K, Sternas L, Zaki M, Palumbo A. Pomalidomide plus low-dose dexamethasone in patients with relapsed/refractory multiple myeloma and moderate renal impairment: a pooled analysis of three clinical trials. Leuk Lymphoma. 2016 Dec;57(12):2833-2838. doi: 10.1080/10428194.2016.1177181. Epub 2016 Jun 7. PMID 27267105

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 112 sites: 4 in Austria, 7 in Belgium, 3 in Denmark, 1 in Estonia, 2 in Finland, 13 in France, 17 in Germany, 1 in Greece, 3 in Ireland, 15 in Italy, 5 in the Netherlands, 2 in Norway, 3 in Poland, 4 in Portugal, 1 in Slovakia, 15 in Spain, 2 in Sweden, 3 in Switzerland, 2 in Turkey, and 9 in the United Kingdom.
Pre-assignment Details: Study participants had to have either refractory or relapsed and refractory disease, defined as documented disease progression during or within 60 days of completing their last myeloma therapy to be eligible to participate in the trial.
Groups:
- Pomalidomide Plus Low Dose Dexamethasone (LD-Dex): Participants received 4 mg pomalidomide (POM) by mouth (PO) on Days 1 to 21 of each 28-day treatment cycle and low dose dexamethasone (LD-Dex) PO at the starting dose of 40 mg/day (≤ 75 years old) or 20 mg/day (> 75 years old) on Days 1, 8, 15 and 22 of a 28-day cycle until the documentation of confirmed progressive disease (PD), intolerable toxicity, death, withdrawal of participation in the study/consent, lost to follow-up, or as long as they benefited from therapy according to the opinion of the responsible study investigator.
Period: Overall Study
Arm/Group | Pomalidomide Plus Low Dose Dexamethasone (LD-Dex)
Started | 682
Received Study Treatment | 676
Completed (Completed = did not discontinue treatment Note: "Reason for Not Completed" below equates to "Reason for Treatment Discontinuation") | 0
Not Completed | 682
Not completed — Lack of Efficacy | 2
Not completed — Lost to Follow-up | 1
Not completed — Progressive Disease | 504
Not completed — Death | 57
Not completed — Adverse Event | 52
Not completed — Miscellaneous | 31
Not completed — Withdrawal by Subject | 21
Not completed — Transition to Commercial Treatment | 8
Not completed — Participants Did Not Receive Study Drug | 6

BASELINE CHARACTERISTICS:
Population: The intent to treat (ITT) population was defined as all enrolled participants (participants who received an interactive voice response system (IVRS) enrollment date) regardless of whether they received any investigational product (IP) or not.
Arm/Group | Pomalidomide Plus Low Dose Dexamethasone (LD-Dex)
Number analyzed (Participants) | 682
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.4 (9.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 301
  Male | 381
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 52
  Not Hispanic or Latino | 626
  Unknown or Not Reported | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 3
  Black or African American | 4
  White | 669
  Other | 2
  Missing | 4
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — ECOG performance status is used to describe a patient's level of functioning in terms of their ability to care for themselves, daily activity, and physical ability (walking, working, etc.). The scale ranges from 0 to 5: 0 = Fully active, no restrictions; 1 = Restricted activity but ambulatory, able to carry out work of a light nature; 2 = Ambulatory and capable of all self-care but unable to carry out work activities; 3 = Limited self-care, confined to bed or chair more than 50% of waking hours; 4 = Completely disabled, no self-care, confined to bed or chair; 5 = Dead
  Participants
    0 = Fully active, no restrictions | 295
    1 = Restricted activity but ambulatory | 319
    2 = Ambulatory and capable of all self-care | 67
    3 = Limited self-care | 1
    4 = Completely disabled | 0
Time since diagnosis [Mean (Standard Deviation); unit: Years] | 6.15 (3.649)
Beta 2 Microglobulin [Mean (Standard Deviation); unit: mg/L] — This test measures the amount of a protein called beta-2 microglobulin (B2M) in the blood.
  mg/L | 5.48 (4.713)
Serum Light Chain Type [Count of Participants; unit: Participants] — Light chains are proteins made by plasma cells and make immunoglobulins (antibodies). Immunoglobulins help protect the body against illness and infections. Immunoglobulins are formed when light chains link up with heavy chains, another type of protein. There are two types of light chains: lambda and kappa light chains. A free light chains test measures the amount of lambda and kappa free light chains in the blood. If the amount of free light chains is higher or lower than normal, it can mean you have a disorder of the plasma cells.
  Participants
    Kappa | 364
    Lambda | 230
    No Serum Light chain Type Detected | 16
    Test Not Performed | 72
Serum Heavy Chain Type [Count of Participants; unit: Participants] — Immunoglobulins help protect the body against illness and infections. Immunoglobulins are formed when light chains link up with heavy chains, another type of protein.
  Participants
    Immunoglobulin A (IgA) | 145
    Immunoglobulin D (IgD) | 5
    Immunoglobulin E (IgE) | 0
    Immunoglobulin G (IgG) | 388
    Immunoglobulin M (IgM) | 4
    No serum heavy chain type detected | 68
    Test not performed | 72
Renal Function (Cockcroft Gault Creatinine Clearance) [Count of Participants; unit: Participants]
  < 30 mL/min | 12
  30 - < 45 mL/min | 57
  45 - < 60 mL/min | 168
  60 - < 80 mL/min | 190
  ≥ 80 mL/min | 250
  Missing | 5
Corrected Serum Calcium [Mean (Standard Deviation); unit: mmol/L] | 2.43 (0.231)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAE)
Description: An adverse event (AE) is any noxious, unintended, or untoward medical occurrence that may appear or worsen in a subject during the course of a study. It may be a new intercurrent illness, a worsening concomitant illness, an injury, or any concomitant impairment of the subject's health, regardless of etiology. Any worsening (i.e., any significant adverse change in the frequency or intensity of a pre- existing condition) was considered an AE. The severity of AEs were graded based on the symptoms according to version 4.0 of the National Cancer Institute Common Terminology Criteria for Adverse Events. Second primary malignancies were monitored as events of interest and considered as part of the assessment of AEs.
  A SAE = AE occurring at any dose that:
  * Results in death;
  * Is life-threatening
  * Requires inpatient hospitalization or prolongation of existing hospitalization
  * Results in persistent or significant disability/incapacity
  * Is a congenital anomaly/birth defect
Time Frame: From the first dose of study treatment up to 28 days following the last dose of study treatment. The median duration of treatment with pomalidomide and LD-dex was 21.4 weeks.
Population: The safety population includes all enrolled participants who received at least one dose of the IP.
Measure: Count of Participants; unit: Participants
Arm/Group | Pomalidomide Plus Low Dose Dexamethasone (LD-Dex)
Number analyzed (Participants) | 676
Participants
  ≥ TEAE | 673
  ≥ 1 TEAE Related to Pomalidomide (POM) | 527
  ≥ 1 TEAE Related to LD-Dex | 448
  ≥ 1 TEAE Related to Either POM or LD-Dex | 575
  ≥ 1 Grade (Gr) 3 or 4 TEAE | 606
  ≥ 1 Gr 3 or 4 TEAE Related to (R/T) POM | 417
  ≥ 1 Gr 3 or 4 TEAE R/T LD-Dex | 226
  ≥ 1 Gr 3 or 4 TEAE R/T Either POM or LD-Dex | 448
  ≥ 1 Grade 5 TEAE | 127
  ≥ 1 Grade 5 TEAE R/T POM | 14
  ≥ 1 Grade 5 TEAE R/T LD-Dex | 16
  ≥ 1 Grade 5 TEAE R/T either POM or LD-Dex | 18
  ≥ 1 Serious TEAE | 448
  ≥ 1 Serious TEAE R/T POM | 187
  ≥ 1 Serious TEAE R/T LD-Dex | 146
  ≥ 1 Serious TEAE R/T Either POM or LD-Dex | 215
  ≥ 1 Serious TEAE Leading to (L/T)Stopping of POM | 36
  ≥ 1 Serious TEAE L/T Stopping of LD-Dex | 34
  ≥1 Serious TEAE L/T Stopping either POM or LD-Dex | 37
  ≥ 1 TEAE L/T to Stopping of POM | 54
  ≥ 1 TEAE L/T to Stopping of LD-DEX | 61
  ≥ 1 TEAE L/T to Stopping of Either POM or LD-DEX | 63
  ≥1 Study Drug Related TEAE (L/T) Stopping POM | 30
  ≥1 Study Drug Related TEAE L/T Stopping LD-Dex | 19
  ≥1 Drug Related TEAE L/T Stopping LD-Dex or POM | 38
  ≥ 1 TEAE L/T to Reduction (R/D) of POM | 164
  ≥ 1 TEAE L/T to R/D of LD-DEX | 150
  ≥ 1 TEAE L/T to R/D of Either POM or LD-DEX | 244
  ≥ 1 Study Drug Related TEAE L/T to R/D of POM | 142
  ≥ 1 Study Drug Related TEAE L/T to R/D of LD-DEX | 135
  ≥1 StudyDrug Related TEAE L/T to R/D POM or LD-DEX | 224
  ≥ 1 TEAE L/T to Interruption (I/R) of POM | 455
  ≥ 1 TEAE L/T to I/R of LD-DEX | 434
  ≥ 1 TEAE L/T to I/R of either POM or LD-DEX | 470
  ≥ 1 Study Drug Related TEAE L/T to I/R of POM | 294
  ≥ 1 Study Drug Related TEAE L/T to I/R of LD-DEX | 185
  ≥1 StudyDrug Related TEAE L/T to I/R POM or LD-DEX | 333

2. Secondary Outcome: Overall Response
Description: Overall response rate (ORR) was defined as the percentage of participants with a stringent complete response (sCR), complete response (CR), very good partial response (VGPR) or partial response (PR) according to the International Myeloma Working Group uniform response criteria (IMWG URC) assessed by the Investigator. Responses must have been confirmed at at least 2 consecutive assessments before the institution of any new therapy with no known evidence of progressive or new bone lesions
Time Frame: Response was assessed at each treatment cycle and at treatment discontinuation; median duration of treatment with pomalidomide and LD-dex was 21.4 weeks
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pomalidomide Plus Low Dose Dexamethasone (LD-Dex)
Number analyzed (Participants) | 682
Percentage of Participants | 33.4 [29.9 to 37.1]

3. Secondary Outcome: Time to Response
Description: Time to response was defined as the time from treatment enrollment to the first documentation of response (sCR, CR, VGPR or PR) based on IMWG criteria.
Time Frame: as for outcome 2
Population: Includes participants with a response (sCR, VGPR or PR).
Measure: Median (Full Range); unit: Weeks
Arm/Group | Pomalidomide Plus Low Dose Dexamethasone (LD-Dex)
Number analyzed (Participants) | 228
Weeks | 8.1 [2 to 112]

4. Secondary Outcome: Kaplan Meier Estimate of Duration of Response
Description: Duration of response, calculated for responders only, was defined as time from the initial documented response (SCR, CR, VGPR or PR) to the first confirmed disease progression, or death if no disease progression was recorded. Participants without a documented progression were censored at the time of their last tumor assessment.
Time Frame: From enrollment to the end of follow-up; median time on follow-up was 10.9 (range 0 - 81) months
Population: Includes participants with a response (sCR, VGPR or PR).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pomalidomide Plus Low Dose Dexamethasone (LD-Dex)
Number analyzed (Participants) | 228
Months | 7.9 [6.48 to 8.78]

5. Secondary Outcome: Kaplan Meier Estimate of Progression Free Survival (PFS) According to the European Medicines Agency Guidelines
Description: Progression free survival was calculated as the time from study enrollment, defined as the IVRS enrollment date, until either PD or death (any cause). Participants without an event (either a documented PD or death) at the time of study end were censored at the time of their last documented disease assessment or at the IVRS enrollment date if no disease assessment was conducted.
Time Frame: From enrollment to the end of follow-up; median time on follow-up was 10.9 (range 0 - 81) months
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pomalidomide Plus Low Dose Dexamethasone (LD-Dex)
Number analyzed (Participants) | 682
Months | 4.6 [3.91 to 4.90]

6. Secondary Outcome: Kaplan Meier Estimate of Time to Progression
Description: Time to progression was calculated as the time from study enrollment until first recorded disease progression as determined by the site investigator based on the IMWG criteria, or until death due to progression. Participants not experiencing a documented progression were censored at the time of their last tumor assessment (or at the time of trial enrollment if no assessment was conducted).
Time Frame: From enrollment to the end of follow-up; median time on follow-up was 10.9 (range 0 - 81) months
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pomalidomide Plus Low Dose Dexamethasone (LD-Dex)
Number analyzed (Participants) | 682
Months | 4.8 [4.27 to 5.56]

7. Secondary Outcome: Kaplan Meier Estimate of Overall Survival (OS)
Description: Overall survival was calculated as the time from study enrollment, defined as the IVRS enrollment date, until death due to any cause. Participants who did not have death data at the time of study end/analysis were censored at the time they were last known to be alive.
Time Frame: From enrollment to the end of follow-up; median time on follow-up was 10.9 (range 0 - 81) months
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pomalidomide Plus Low Dose Dexamethasone (LD-Dex)
Number analyzed (Participants) | 682
Months | 11.9 [10.65 to 13.41]

8. Secondary Outcome: Pomalidomide Exposure - Apparent (Oral) Clearance (CL/F)
Description: Pharmacokinetic (PK) parameters are derived from pomalidomide concentration versus time data.
Time Frame: Cycles 1, 2, 3, 4, 5, 6
Population: Pharmacokinetic population
  Pharmacokinetic samples from 476 participants included in studies CC-4047-MM-005 and CC 4047 MM 010 were used for the population PK analysis of pomalidomide
Measure: Median (95% Confidence Interval); unit: Liters/hour
Arm/Group | Pomalidomide Plus Low Dose Dexamethasone (LD-Dex)
Number analyzed (Participants) | 476
Liters/hour | 6.02 [5.67 to 6.48]

9. Secondary Outcome: Pomalidomide Exposure - Apparent Volume of Distribution (V/F)
Description: Pharmacokinetic (PK) parameters are derived from Pomalidomide concentration versus time data.
Time Frame: Cycles 1, 2, 3, 4, 5, 6
Population: as for outcome 8
Measure: Median (95% Confidence Interval); unit: Liters
Arm/Group | Pomalidomide Plus Low Dose Dexamethasone (LD-Dex)
Number analyzed (Participants) | 476
Liters | 75.10 [63.57 to 89.17]

10. Secondary Outcome: Cytogenetic Analysis
Description: Cytogenetic analysis was to be performed using fluorescence in situ hybridization (FISH) methodology at a local laboratory, to evaluate the relationship between cytogenetic profiles and the combination of POM and LD-DEX in terms of response and outcome.
Time Frame: Study entry
Population: Statistical analysis could not be performed due to high level of missing cytogenetic data as well as cytogenetic probe analysis being non- compliant with study requirements which lead to an inability to accurately identify specific cytogenetic abnormalities.
Arm/Group | Pomalidomide Plus Low Dose Dexamethasone (LD-Dex)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: All-cause mortality is reported from enrollment until the end of follow-up; median time on follow-up was 10.9 (range 0 - 81) months. Adverse events are reported from first dose of study drug up to 28 days after last dose; median duration of treatment was 21.4 weeks.
Description: Second primary malignancies were monitored as events of interest and considered as part of the assessment of AEs.
Arm/Group | Pomalidomide Plus Low Dose Dexamethasone (LD-Dex)
All-Cause Mortality (participants affected / at risk) | 598/682
Serious Adverse Events (participants affected / at risk) | 448/676
Other Adverse Events (participants affected / at risk) | 646/676
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pomalidomide Plus Low Dose Dexamethasone (LD-Dex) (N=676)
Anaemia (Blood and lymphatic system disorders) | 15
Bone marrow failure (Blood and lymphatic system disorders) | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 34
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 1
Hyperviscosity syndrome (Blood and lymphatic system disorders) | 3
Leukopenia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 20
Pancytopenia (Blood and lymphatic system disorders) | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 13
Acute coronary syndrome (Cardiac disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 1
Angina pectoris (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 17
Atrial flutter (Cardiac disorders) | 3
Atrioventricular block (Cardiac disorders) | 1
Cardiac amyloidosis (Cardiac disorders) | 2
Cardiac arrest (Cardiac disorders) | 2
Cardiac disorder (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 12
Cardiac failure congestive (Cardiac disorders) | 2
Cardio-respiratory arrest (Cardiac disorders) | 2
Coronary artery stenosis (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 4
Nodal arrhythmia (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 1
Sinus bradycardia (Cardiac disorders) | 1
Conjunctival haemorrhage (Eye disorders) | 1
Exophthalmos (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 3
Abdominal pain upper (Gastrointestinal disorders) | 2
Anal fistula (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 6
Diverticulum intestinal (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 2
Gastrointestinal amyloidosis (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Intestinal infarction (Gastrointestinal disorders) | 1
Large intestinal haemorrhage (Gastrointestinal disorders) | 1
Large intestine perforation (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Pancreatitis (Gastrointestinal disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1
Rectal ulcer (Gastrointestinal disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Volvulus (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 4
Asthenia (General disorders) | 5
Death (General disorders) | 4
Disease progression (General disorders) | 1
Euthanasia (General disorders) | 1
Fatigue (General disorders) | 5
General physical health deterioration (General disorders) | 45
Generalised oedema (General disorders) | 1
Hyperpyrexia (General disorders) | 2
Hyperthermia (General disorders) | 1
Malaise (General disorders) | 2
Mucosal inflammation (General disorders) | 1
Multiple organ dysfunction syndrome (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Oedema (General disorders) | 1
Oedema peripheral (General disorders) | 2
Pain (General disorders) | 2
Pyrexia (General disorders) | 41
Cholecystitis (Hepatobiliary disorders) | 1
Cholecystitis acute (Hepatobiliary disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Gallbladder obstruction (Hepatobiliary disorders) | 1
Hepatic failure (Hepatobiliary disorders) | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1
Liver disorder (Hepatobiliary disorders) | 1
Drug hypersensitivity (Immune system disorders) | 1
Abdominal infection (Infections and infestations) | 1
Abscess limb (Infections and infestations) | 1
Anal abscess (Infections and infestations) | 1
Appendicitis (Infections and infestations) | 1
Arthritis bacterial (Infections and infestations) | 1
Atypical pneumonia (Infections and infestations) | 4
Bacteraemia (Infections and infestations) | 2
Bacterial diarrhoea (Infections and infestations) | 1
Biliary sepsis (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 9
Bronchopulmonary aspergillosis (Infections and infestations) | 4
Bursitis infective (Infections and infestations) | 1
Campylobacter gastroenteritis (Infections and infestations) | 1
Catheter site infection (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 2
Cerebral aspergillosis (Infections and infestations) | 1
Citrobacter infection (Infections and infestations) | 1
Clostridial sepsis (Infections and infestations) | 1
Clostridium difficile colitis (Infections and infestations) | 2
Cystitis (Infections and infestations) | 1
Device related infection (Infections and infestations) | 2
Diverticulitis (Infections and infestations) | 2
Ear infection (Infections and infestations) | 1
Erysipelas (Infections and infestations) | 1
Escherichia infection (Infections and infestations) | 1
Escherichia sepsis (Infections and infestations) | 4
Escherichia urinary tract infection (Infections and infestations) | 1
Folliculitis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 5
Gastroenteritis norovirus (Infections and infestations) | 1
Herpes zoster infection neurological (Infections and infestations) | 1
Infection (Infections and infestations) | 14
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1
Influenza (Infections and infestations) | 5
Leishmaniasis (Infections and infestations) | 1
Listeria sepsis (Infections and infestations) | 1
Listeriosis (Infections and infestations) | 1
Localised infection (Infections and infestations) | 1
Lower respiratory tract infection (Infections and infestations) | 22
Lung infection (Infections and infestations) | 16
Meningitis pneumococcal (Infections and infestations) | 1
Meningococcal sepsis (Infections and infestations) | 1
Neutropenic sepsis (Infections and infestations) | 5
Oral fungal infection (Infections and infestations) | 1
Oral infection (Infections and infestations) | 1
Osteomyelitis bacterial (Infections and infestations) | 1
Otitis externa (Infections and infestations) | 1
Parainfluenzae virus infection (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Pneumococcal sepsis (Infections and infestations) | 1
Pneumocystis jirovecii pneumonia (Infections and infestations) | 3
Pneumonia (Infections and infestations) | 117
Pneumonia influenzal (Infections and infestations) | 3
Pneumonia pneumococcal (Infections and infestations) | 5
Pneumonia respiratory syncytial viral (Infections and infestations) | 2
Pneumonia staphylococcal (Infections and infestations) | 2
Pneumonia streptococcal (Infections and infestations) | 2
Pneumonia viral (Infections and infestations) | 1
Pseudomonal sepsis (Infections and infestations) | 3
Pulmonary sepsis (Infections and infestations) | 3
Respiratory moniliasis (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 11
Rhinovirus infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 14
Septic shock (Infections and infestations) | 15
Sinusitis bacterial (Infections and infestations) | 1
Soft tissue infection (Infections and infestations) | 1
Staphylococcal infection (Infections and infestations) | 1
Staphylococcal sepsis (Infections and infestations) | 3
Staphylococcal skin infection (Infections and infestations) | 1
Streptococcal bacteraemia (Infections and infestations) | 1
Streptococcal infection (Infections and infestations) | 2
Systemic candida (Infections and infestations) | 1
Systemic infection (Infections and infestations) | 1
Tracheobronchitis (Infections and infestations) | 2
Upper respiratory tract infection (Infections and infestations) | 8
Urinary tract infection (Infections and infestations) | 11
Urinary tract infection bacterial (Infections and infestations) | 1
Urosepsis (Infections and infestations) | 5
Vascular device infection (Infections and infestations) | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 3
Febrile nonhaemolytic transfusion reaction (Injury, poisoning and procedural complications) | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 2
Femur fracture (Injury, poisoning and procedural complications) | 4
Head injury (Injury, poisoning and procedural complications) | 1
Humerus fracture (Injury, poisoning and procedural complications) | 4
Ilium fracture (Injury, poisoning and procedural complications) | 2
Joint dislocation (Injury, poisoning and procedural complications) | 1
Perineal injury (Injury, poisoning and procedural complications) | 1
Post-traumatic pain (Injury, poisoning and procedural complications) | 1
Rib fracture (Injury, poisoning and procedural complications) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1
Traumatic fracture (Injury, poisoning and procedural complications) | 1
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 1
Blood creatinine increased (Investigations) | 6
Blood immunoglobulin A increased (Investigations) | 1
C-reactive protein increased (Investigations) | 2
International normalised ratio increased (Investigations) | 1
Monoclonal immunoglobulin present (Investigations) | 3
Neutrophil count decreased (Investigations) | 2
Platelet count decreased (Investigations) | 1
Protein urine present (Investigations) | 1
White blood cell count decreased (Investigations) | 2
Decreased appetite (Metabolism and nutrition disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 5
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1
Hyperamylasaemia (Metabolism and nutrition disorders) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 30
Hyperglycaemia (Metabolism and nutrition disorders) | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 2
Metabolic acidosis (Metabolism and nutrition disorders) | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 7
Bone lesion (Musculoskeletal and connective tissue disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 7
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 2
Osteolysis (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Pathological fracture (Musculoskeletal and connective tissue disorders) | 7
Spinal pain (Musculoskeletal and connective tissue disorders) | 4
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Monoclonal gammopathy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Plasma cell leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Cauda equina syndrome (Nervous system disorders) | 1
Cerebral haematoma (Nervous system disorders) | 1
Cognitive disorder (Nervous system disorders) | 1
Coma (Nervous system disorders) | 1
Depressed level of consciousness (Nervous system disorders) | 2
Disturbance in attention (Nervous system disorders) | 1
Encephalopathy (Nervous system disorders) | 1
Facial nerve disorder (Nervous system disorders) | 1
Generalised tonic-clonic seizure (Nervous system disorders) | 1
Haemorrhage intracranial (Nervous system disorders) | 2
Headache (Nervous system disorders) | 1
IIIrd nerve paresis (Nervous system disorders) | 1
Intracranial aneurysm (Nervous system disorders) | 1
Lateral medullary syndrome (Nervous system disorders) | 1
Motor dysfunction (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Paraplegia (Nervous system disorders) | 1
Parkinsonism (Nervous system disorders) | 1
Peripheral motor neuropathy (Nervous system disorders) | 1
Peripheral sensorimotor neuropathy (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 1
Ruptured cerebral aneurysm (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 2
Somnolence (Nervous system disorders) | 1
Spinal cord compression (Nervous system disorders) | 3
Subarachnoid haemorrhage (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 2
Confusional state (Psychiatric disorders) | 4
Depression (Psychiatric disorders) | 1
Disorientation (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 26
Crush syndrome (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Oliguria (Renal and urinary disorders) | 2
Renal failure (Renal and urinary disorders) | 23
Renal impairment (Renal and urinary disorders) | 1
Renal vascular thrombosis (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Scrotal cyst (Reproductive system and breast disorders) | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 15
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 5
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 14
Rash (Skin and subcutaneous tissue disorders) | 1
Skin necrosis (Skin and subcutaneous tissue disorders) | 1
Social stay hospitalisation (Social circumstances) | 1
Aortic stenosis (Vascular disorders) | 1
Deep vein thrombosis (Vascular disorders) | 6
Haematoma (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 4
Shock haemorrhagic (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pomalidomide Plus Low Dose Dexamethasone (LD-Dex) (N=676)
Anaemia (Blood and lymphatic system disorders) | 327
Leukopenia (Blood and lymphatic system disorders) | 92
Neutropenia (Blood and lymphatic system disorders) | 382
Thrombocytopenia (Blood and lymphatic system disorders) | 236
Abdominal pain (Gastrointestinal disorders) | 34
Constipation (Gastrointestinal disorders) | 163
Diarrhoea (Gastrointestinal disorders) | 118
Nausea (Gastrointestinal disorders) | 96
Vomiting (Gastrointestinal disorders) | 49
Asthenia (General disorders) | 155
Fatigue (General disorders) | 197
Oedema peripheral (General disorders) | 108
Pyrexia (General disorders) | 178
Bronchitis (Infections and infestations) | 70
Nasopharyngitis (Infections and infestations) | 57
Pneumonia (Infections and infestations) | 38
Respiratory tract infection (Infections and infestations) | 58
Upper respiratory tract infection (Infections and infestations) | 50
Urinary tract infection (Infections and infestations) | 54
Blood creatinine increased (Investigations) | 49
C-reactive protein increased (Investigations) | 34
Neutrophil count decreased (Investigations) | 47
Weight decreased (Investigations) | 47
Decreased appetite (Metabolism and nutrition disorders) | 69
Hypercalcaemia (Metabolism and nutrition disorders) | 40
Hyperglycaemia (Metabolism and nutrition disorders) | 40
Hypokalaemia (Metabolism and nutrition disorders) | 52
Arthralgia (Musculoskeletal and connective tissue disorders) | 42
Back pain (Musculoskeletal and connective tissue disorders) | 105
Bone pain (Musculoskeletal and connective tissue disorders) | 65
Muscle spasms (Musculoskeletal and connective tissue disorders) | 96
Muscular weakness (Musculoskeletal and connective tissue disorders) | 35
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 54
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 37
Pain in extremity (Musculoskeletal and connective tissue disorders) | 54
Dizziness (Nervous system disorders) | 55
Headache (Nervous system disorders) | 49
Peripheral sensory neuropathy (Nervous system disorders) | 79
Tremor (Nervous system disorders) | 45
Confusional state (Psychiatric disorders) | 37
Insomnia (Psychiatric disorders) | 76
Cough (Respiratory, thoracic and mediastinal disorders) | 141
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 117
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 47
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 37
Pruritus (Skin and subcutaneous tissue disorders) | 36
Rash (Skin and subcutaneous tissue disorders) | 54

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Results from a center cannot be submitted for publication before results of multicenter study are published unless it is > 1 year since study completion. Then, Investigator can publish if manuscript is submitted to Celgene 60 days prior to submission. If Celgene decides publication would hinder drug development, Investigator must delay submission for up to 90 additional days. Investigator must delete confidential information before submission and defer publication to permit patent applications.

DOCUMENTS (2):
  • Study Protocol (2013-05-30): https://cdn.clinicaltrials.gov/large-docs/89/NCT01712789/Prot_000.pdf
  • Statistical Analysis Plan (2015-03-06): https://cdn.clinicaltrials.gov/large-docs/89/NCT01712789/SAP_001.pdf